CLINICAL TRIAL: NCT06310837
Title: Effect of Immunosuppressants With Adalimumab Biosimilars vs Corticosteroids on Noninfectious Uveitis: A Multicenter, Randomized, Non-inferiority Clinical Trial
Brief Title: Effect of Immunosuppressants With Adalimumab Biosimilars vs Corticosteroids on Noninfectious Uveitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: The Eye Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Shandong Eye Hospital (Other); Shenzhen Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KYPJ300
Record Dates: First submitted 2024-02-20; First posted 2024-03-15 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Uveitis
Keywords: Uveitis; Corticosteroids; Adalimumab biosimilars
MeSH Terms: conditions — Uveitis | interventions — Adrenal Cortex Hormones; Immunosuppressive Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADA+MMF group (Experimental): Adalimumab biosimilars with immunosuppressants therapy
  Interventions: Drug: Adalimumab Biosimilars Injection; Drug: Immunosuppressive Agents
- Corticosteroids+MMF group (Active Comparator): Corticosteroids with immunosuppressive therapy；
  Interventions: Drug: Corticosteroid; Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Adalimumab Biosimilars Injection — Adalimumab biosimilars: 80 mg was subcutaneously injected for the first time in the first week, and then 40 mg was subcutaneously injected every two weeks from the first week to the 48 th week.
  Other Names: Subcutaneous injection of adalimumab biosimilars
  Arms: ADA+MMF group
Drug: Corticosteroid — Patients received no less than 1 mg / kg.d glucocorticoid at week 0, then implemented according to the standard reduction scheme.
  Other Names: Oral corticosteroids
  Arms: Corticosteroids+MMF group
Drug: Immunosuppressive Agents — Mycophenolate mofetil 1g bid for more than 3 months, maintenance dose not less than 0.5g bid
  Other Names: Immunosuppressant

SUMMARY:
This is a multi-center, prospective, randomized controlled non-inferior clinical study. A total of 120 subjects with non-infectious intermediate, posterior, or panuveitis were enrolled in Zhongshan Ophthalmic Center and three other centers. They were randomly assigned to the experimental group and the control group according to ( 1 : 1 ). We hypothesized that adalimumab biosimilars combined with immunosuppressive agents in the treatment of non-infectious uveitis is not inferior to glucocorticoids combined with immunosuppressive agents, and there are no additional adverse events and safety issues.

DETAILED DESCRIPTION:
The study will be followed up in the screening-baseline period and at 4,8,12,18,24,36, and 48 weeks after the start of the study drug. The ETDRS letter number change of the best corrected visual acuity ( BCVA ) at 24 weeks compared with the baseline was used as the main indicator. The last follow-up was performed at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old ( including boundary value ), male or female.
2. At least one eye is diagnosed as noninfectious intermediate uveitis, posterior uveitis or panuveitis.
3. Subject is on prednisone ≥ 10 mg/day (or corticosteroid equivalent) for at least 2 weeks prior to Screening and remains on the same dose from screening to baseline visit.
4. At least one eye is diagnosed as active uveitis at baseline；
5. Subject is voluntary to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Subject with isolated anterior uveitis.
2. Subject with prior inadequate response to or intolerance to high-dose corticosteroids (equivalent of prednisone 1 mg/kg/day or 60 to 80 mg/day).
3. Subject is suspected or diagnosed as infectious uveitis.
4. Uncontrolled glaucoma or high intraocular pressure, defined as intraocular pressure>25 mmHg after treatment with ≥ 2 anti-glaucoma drugs or evidence of glaucomatous optic nerve injury.
5. Subject with best corrected visual acuity (BCVA) worse than 20/400 (ETDRS logMAR > 1.34 or <20 letters) in the better eye.
6. Subject with other fundus diseases.
7. Subject with demyelinating diseases.
8. Subject has a contraindication to pupil dilation with mydriatic eyedrops.
9. Subject with corneal or lens opacity that precludes visualization of the anterior segment and fundus.
10. Topical corticosteroids and/or topical NSAID>3 drops per day in the 14 days prior to baseline; Dexamethasone/betamethasone or equivalent subconjunctival steroid within 30 days prior to baseline; Parafbulbar, intravitreal (IVT), suprasoroidal, or periocular corticosteroid injections were administered within 60 days prior to baseline; Received IVT anti-VEGF therapies less than 60 days prior to baseline; Dexamethasone (Ozurdex) IVT implant within 6 months prior to baseline; Fluocinolone acetonide IVT implant within 3 years prior to baseline.
11. Subject with history of prior intraocular surgery within 90 days prior to baseline or any planned (elective) eye surgery within the next 1 year from baseline.
12. Subject is diagnosised or suspected tuberculosis, hepatitis B virus, hepatitis C virus, HIV, syphilis infection or with other uncontrolled active infections or other infections that would put the subject at uncontrolled risk.
13. Subject with severe, progressive, or uncontrolled symptoms of renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiovascular, neurological, or cerebral diseases or with malignant tumors or with moderate to severe heart failure and subjects who are considered by the investigator to be at unacceptable risk by participating in the study.
14. Prior biologic and immunosuppressant therapy other than corticosteroids at any time.
15. Subject with a systemic inflammatory disease that requires continued therapy with oral corticosteroids or a prohibited immunosuppressive agent at Screening or Baseline visits.
16. Fertile woman who has a positive serum pregnancy test at the screening visit or plans for pregnancy and sperm donation during the trial and within 6 months after the end of the study.
17. Other subjects who are considered by the investigator to be inappropriated for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of ETDRS letter count for BCVA at week 24 from baseline | week 24
  The best corrected visual acuity of the patient would be examined by the ETDRS visual acuity chart according to the visual acuity examination SOP. Change of ETDRS letter count for BCVA at week 24 from baseline were the main indicator, the outcome at other follow-up time points（Baseline, weeks 4, 8, 12, 18, 36, 48）would also be included in the outcome analysis.

SECONDARY OUTCOMES:
Proportion of patients with weight gain at week 24 from baseline | week 24
  Patients would be instructed to remove shoes and heavy clothing for measurement, and weight gain is defined as a 5% increase from baseline.
Time of treatment failures | week 24
  Treatment failure is defined as an increase in the degree of inflammation in one or more of four areas, including choroidal and/or retinal vasculopathy, macular edema, anterior chamber cell grade, and vitreous opacity grade, assessed by the investigators from week 4 to the end of follow-up.
Number of treatment failures | week 24
  Treatment failure is defined as an increase in the degree of inflammation in one or more of four areas, including choroidal and/or retinal vasculopathy, macular edema, anterior chamber cell grade, and vitreous opacity grade, assessed by the investigators from week 4 to the end of follow-up.
Change of Visual Functioning Questionnaire- 25 (VFQ-25) composite score from baseline | week 24
  The changes of each follow-up time point from the baseline are evaluated according to VFQ-25 visual function evaluation scale.To calculate an overall composite score for the VFQ-25, we will simply average the vision-targeted subscale scores, excluding the general health rating question.(100=best, 0=worst possible score)
Change of anterior chamber inflammation at week 24 from baseline | week 24
  Change of anterior chamber inflammation assessed by research doctors with slit-lamp according to the International Uveitis Organization ( SUN group ) classification criteria.
Change of vitreous opacity at week 24 from baseline | week 24
  Change of vitreous opacity assessed by research doctors with slit-lamp according to the International Uveitis Organization ( SUN group ) classification criteria.
Change of the retinal and choroidal inflammation at week 24 from baseline | week 24
  Change of the retinal and choroidal inflammation assessed by fluorescein angiography.
Change of the thickness of retina and choroid in macular area at week 24 from baseline | week 24
  Change of the thickness of retina and choroid in macular area evaluated by Optical Coherence Tomography (OCT) or Optical Coherence Tomography Angiography (OCTA).
Occurrence of skin abnormalities at the end of study | week 48
  The occurrence of skin abnormalities reported by research doctors based on adverse reaction evaluation criteria (CTCAE v5.0).
Occurrence of hypertension at the end of study | week 48
  The occurrence of hypertension assessed by electronic blood manometer based on adverse reaction evaluation criteria (CTCAE v5.0).
Occurrence of hyperglycemia at the end of study | week 48
  The occurrence of hyperglycemia assessed by venous blood glucose testing based on adverse reaction evaluation criteria (CTCAE v5.0).
Occurrence of active tuberculosis infection at the end of study | week 48
  The occurrence of active tuberculosis infection assessed by pulmonary X-ray examination and tuberculosis bacterial T cell detection and evaluated by research doctors.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chi, Principal Investigator — Shenzhen Eye Hospital
Locations (1):
- Shenzhen Eye Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No